CLINICAL TRIAL: NCT00421356
Title: Kinetic and Kinematic Comparison of Power Assisted Versus Stance Control Artificial Knees During Sit To Stand
Brief Title: Comparison of Prosthetic Knee Performance During Sitting and Standing
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Jason Highsmith, Assistant Professor, University of South Florida
Other Study IDs: 104850; US DOE RSA Award # H235J050020
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Amputation
Keywords: amputation, transfemoral, lower extremity, prosthetic knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Transfemoral Power Knee group: Transfemoral amputees who used the power assisted Ossur Power Knee who used the knee daily without adjustments for at least 90 days prior to the study.
- Transfemoral C-Leg knee group: Transfemoral amputees who used the stance control Otto Bock C-Leg who used the knee daily without adjustments for at least 90 days prior to the study.
- Transfemoral Mauch knee group: Transfemoral amputees who used the mechanical fluid controlled Mauch Swing and Stance Knee who used the knee daily without adjustments for at least 90 days prior to the study.
- Non amputee control group: Healthy, non-amputee control group

SUMMARY:
The Ossur Prosthetic Power Knee claims to assist in helping people with transfemoral amputation to walk up stairs and stand up from sitting. We expect to find that this product has the ability to help unload the sound knee during these tasks. We plan to collect force and motion data while people stand up from a chair. We will compare the data from people using several types of prosthetic knees, including the power knee as well as from people who are not amputees to see what the force and motion contributions are from the different knees evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 7 control subjects with normal lower extremity function: mentally independent adults with intact extremities. These individuals shall have no significant medical history that would impair their ability to perform 3, repeated, sit to stand trials. Exclusionary examples might include history positive for total joint arthroplasty of the hip or knee and significant cardiomyopathy. Control subjects will be non-amputee, generally healthy individuals, mentally capable of providing informed consent. They will have no significant medical history that could be perceived by investigators to hinder the ability to transfer. Anyone not meeting these criteria cannot be a control subject.
* 28 subjects with unilateral amputation at the level of the thigh. 7 each in four groups:

  1. Active Extension Group: Power Knee
  2. Microprocessor Stance Control Group: C-Leg, Rheo, Adaptive
  3. Non-Microprocessor Stance Control Group: Mauch, Catech or other stance control units
  4. Non-Microprocessor and Non-Stance Control units: WASB, polycentrics, pneumatics Each subject must have a prosthesis for which they have had for a minimum of 90 days in its present condition.
* All subjects must be:

  1. at least 21 years of age,
  2. mentally independent, and
  3. able to give informed consent.

Exclusion Criteria:

* Subjects are not candidates if they:

  1. are under 21 years of age
  2. are mentally dependent and unable to provide their own informed consent
  3. have worn the present prosthesis for less than 90 days in the current condition
  4. have bilateral amputation
* Subjects with an amputation are not candidates if they only use a prosthesis for transfers or therapy (K0 or K1 Medicare functional class). They must be independently ambulatory, at some level in the community (Medicare functional class "K2-K4"). They are furthermore not a candidate for this study if they have bilateral amputation (at any level) of the lower extremity as the purpose is to determine sound versus involved side loading, then against control. If all of the latter criteria are satisfied, the final piece is the 90 day prosthetic accommodation period. Candidacy then hinges upon the fact that they are accommodated to their current prosthesis as evident by having worn the current device, unaltered for the 90 days prior to testing.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with Transfemoral Amputation
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2010-09-30 (Actual); Study Completion 2010-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Jason Highsmith, DPT, CP, Principal Investigator — USF School of Physical Therapy & Rehab Sciences
Locations (1):
- University of South Florida, Tampa, Florida, United States